CLINICAL TRIAL: NCT00362414
Title: Safety of Beta-hCG + Erythropoietin in Acute Stroke
Brief Title: Beta-hCG + Erythropoietin in Acute Stroke
Acronym: BETAS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Stem Cell Therapeutics Corp. (Industry); Hoag Memorial Hospital Presbyterian (Other)
Responsible Party: Principal Investigator, Steven C. Cramer, MD, Professor, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS#2005-4800
Record Dates: First submitted 2006-08-09; First posted 2006-08-10 (Estimated); Results first posted 2016-08-29 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-08

CONDITIONS: Acute Stroke
Keywords: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dual Growth Factor (Experimental): All patients received erythropoietin and beta-hCG. This was the only treatment arm in the study, i.e., all enrollees received active therapy.
  Interventions: Drug: Dual Growth Factor

INTERVENTIONS:
Drug: Dual Growth Factor — 10,000 IU Beta-hCG IV on days 1, 3, and 5 of study participation
  30,000 IU Erythropoietin IV on days 7, 8 and 9 of study participation

SUMMARY:
The purpose of this study is to assess the safety of Beta-hCG + Erythropoietin in patients with acute ischemic stroke.

DETAILED DESCRIPTION:
Patients with a new stroke will be evaluated at the University of California Irvine Medical Center (UCIMC), a JCAHO-certified Stroke Center, and at Hoag Memorial Hospital Presbyterian. Standard stroke pathways will be used to identify such patients and to initiate standard of care therapy. Patients potentially eligible for study enrollment will be identified, screened, then consented and enrolled. Those meeting all entry criteria, and no exclusion criteria, will undergo additional baseline testing including brain MRI. A 9-day course of B-E therapy will then begin, always within 48 hours after stroke onset. This therapy will consist of hCG (3 once-daily IM doses at 10,000 IU per dose, one day apart, on days 1, 3 and 5 of study participation), followed by a one day washout period (day 6), followed by Epo (three once-daily i.v. doses at 30,000 IU per dose on days 7, 8, and 9 of study participation). Patients will be examined at several time points during therapy, as well as 6 weeks and 3 months after stroke onset. The primary outcome measures are related to safety, while secondary outcome measures are related to disability, neurological status, and MRI measures.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21-85
2. NIHSS score 6-24 at time of enrollment, ensuring that stroke is neither mild nor devastating
3. Stroke is ischemic in origin, supratentorial, and radiologically confirmed
4. Patient is 24-48 hours from time of stroke onset at time that first dose of B-E therapy is administered. Time of onset is when symptoms began, and stroke occurred during sleep, time of onset is when patient was last seen to be normal.
5. Reasonable expectation of availability to receive the full 9 day B-E therapy course
6. Reasonable expectation that patient will receive standard post-stroke physical, occupational, speech, and cognitive therapy as indicated

Exclusion Criteria:

1. Pre-existing and active major psychiatric or other neurological disease
2. History of significant alcohol or drug abuse in the prior 3 years
3. Serum hemoglobin > 16 g/dL in a male patient or > 14 g/dL in a female patient; or a platelet count > 400,000/mm3 in either a male or female patient
4. Advanced liver, kidney, cardiac, or pulmonary disease; the former will be operationally defined as a serum bilirubin > 4 mg/dL, alkaline phosphatase > 250 U/L, SGOT > 150 U/L, SGPT >150 U/L, or creatinine > 3.5 mg/dL
5. Pregnancy or lactating; note that a negative pregnancy test will be required if the patient is a female in reproductive years, using a test that reliably detects beta-hCG levels > 25 with normal levels being < 8 IU/L.
6. Contraindication to study participation on the basis of any of the following:

   1. Allergy or other contraindication to initiating either beta-hCG or Erythropoietin
   2. Known hypersensitivity to mammalian cell-derived products or hypersensitivity to albumin
   3. A known diagnosis of prostatic cancer; note that prostate specific antigen will be collected for retrospective assessment of safety, but will not be used to ascertain study eligibility
   4. Dysuria of unexplained origin
   5. Uncontrolled hypertension, defined in the context of acute stroke as blood pressure persistently above 220 mm Hg systolic or 120 diastolic despite antihypertensive therapy
7. Current use of either beta-hCG or Erythropoietin
8. Other condition known to elevate beta-hCG, active in the prior 24 months, e.g., choriocarcinoma or germ cell tumor
9. Terminal medical diagnosis consistent with survival < 1 year
10. Known hypercoagulable state, which for the purposes of this study will deficiency of proteins C, S, or antithrombin III; activated protein C resistance; prothrombin gene mutation; or an anti-phospholipid antibody syndrome as based on clinical and laboratory measures.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2006-08; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven C. Cramer, MD, MMSc, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine Medical Center, Orange, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were consented and enrolled from September 2006 to February 2008 in accordance with local Institutional Review Boards at 3 North American sites: University of California Irvine Medical Center (n=11), Hoag Memorial Hospital Presbyterian (n=1), and the Foothills Hospital at University of Calgary (n=3).
Groups:
- Beta-hCG + Erythropoietin: Subjects received a 9-day course of beta-human chorionic gonadotropin (once daily on Days 1, 3, and 5 of study participation) followed by erythropoietin (once daily on Days 7, 8, and 9 of study participation)
Period: Overall Study
Arm/Group | Beta-hCG + Erythropoietin
Started | 15
Completed | 12
Not Completed | 3
Not completed — Death | 2
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Beta-hCG + Erythropoietin
Number analyzed (Participants) | 15
Age, Continuous [Median (Full Range); unit: years] | 72 [23 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12
  Canada | 3
History of Hypertension [Number; unit: participants]
  Yes | 12
  No | 3
History of Hyperlipidemia [Number; unit: participants]
  Yes | 9
  No | 6
History of Diabetes Mellitus [Number; unit: participants]
  Yes | 6
  No | 9
History of Prior Stroke [Number; unit: participants]
  Yes | 5
  No | 10
History of Atrial Fibrillation [Number; unit: participants]
  Yes | 4
  No | 11

OUTCOME MEASURES:

1. Primary Outcome: Safety
Description: Safety through Day 90 was assessed through adverse event reporting, serial examinations, blood testing, and a leg vein Doppler at Day 42. Number of participants who experienced adverse events, had abnormality in serial examinations, blood testing, and a leg vein Doppler at Day 42.
Time Frame: 3 mo
Measure: Number; unit: participants
Groups:
- Dual Growth Factor: All patients received erythropoietin and beta-hCG. This was the only treatment arm in the study, i.e., all enrollees received active therapy.
  Dual Growth Factor: 10,000 IU Beta-hCG IV on days 1, 3, and 5 of study participation
  30,000 IU Erythropoietin IV on days 7, 8 and 9 of study participation
Arm/Group | Dual Growth Factor
Number analyzed (Participants) | 15
participants | 0

2. Primary Outcome: Morbidity
Description: attributable to experimental intervention
Time Frame: 3 mo
Measure: Number; unit: participants
Arm/Group | Dual Growth Factor
Number analyzed (Participants) | 15
participants | 0

3. Primary Outcome: Mortality
Description: attributable to experimental intervention
Time Frame: 3 mo
Measure: Number; unit: participants
Groups:
- Two Growth Factors: double growth factors
Arm/Group | Two Growth Factors
Number analyzed (Participants) | 15
participants | 0

4. Secondary Outcome: Action Research Arm Test
Description: The Action Research Arm Test is a 19 item measure divided into 4 sub-tests (grasp, grip, pinch, and gross arm movement). Performance on each item is rated on a 4-point ordinal scale ranging from: 3: Performs test normally 2: Completes test, but takes abnormally long or has great difficulty 1: Performs test partially 0: Can perform no part of test. Total scores range from 0-57 points, a higher score being better with 57 being considered "normal".
Time Frame: 3 mo
Population: This number (9) is the total # subjects who could complete the test at all study time points; some subjects were unable to complete this test at one of the time points, especially the acute stroke assessment.
Measure: Median (Full Range); unit: Units on a scale
Groups:
- 2 Growth Factors: double growth factors
Arm/Group | 2 Growth Factors
Number analyzed (Participants) | 9
Units on a scale | 23 [0 to 57]

5. Secondary Outcome: Fugl-Meyer Arm Scale
Description: Fugl-Meyer arm scale is a measurement scale of the upper body with three sections being Proximal, Wrist/Hand, and Coordination/Speed. The scores can range from 0-66 with a higher score being better. A score of 66 is considered "normal" with no impairments.
Time Frame: 3 mo
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | 2 Growth Factors
Number analyzed (Participants) | 12
Units on a scale | 32 [2 to 65]

6. Secondary Outcome: Fugl-Meyer Leg Scale
Description: Measure of leg motor impairment with three subsections which are Proximal, Hip/Knee, and Speed/Coordination. The scale ranges from 0-34 with a higher score being better. A score of 34 is considered "normal".
Time Frame: 3 mo.
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | 2 Growth Factors
Number analyzed (Participants) | 10
Units on a scale | 20 [3 to 34]

7. Secondary Outcome: Boston Naming Test
Description: Measure of aphasia or other language disturbance caused by stroke or other dementing disorders. It consists of 60 line drawings graded in difficulty in which patients are to name each picture.
Time Frame: 3 mo
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | 2 Growth Factors
Number analyzed (Participants) | 13
Units on a scale | 2 [0 to 10]

8. Secondary Outcome: Line Cancellation Test
Description: Measure of spatial neglect where patients must cross out lines placed in a random orientation. Missed lines may indicate areas of spatial neglect.
Time Frame: 3 mo
Measure: Median (Full Range); unit: ratio of canceled lines on each side
Arm/Group | 2 Growth Factors
Number analyzed (Participants) | 8
ratio of canceled lines on each side | 96 [20 to 100]

9. Secondary Outcome: NIH Stroke Scale
Description: Measure of global impairment post stroke. It includes 11 items to examine levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss. The scoring scale is between 0-42 where a higher score is indicative of a more severe stroke.
Time Frame: 3 mo
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | 2 Growth Factors
Number analyzed (Participants) | 15
Units on a scale | 10 [6 to 19]

10. Secondary Outcome: Geriatric Depression Scale Short Form
Description: Measure of depression done as a self-report. It is a series of 15 questions designed to be a screen for depression. The scores range from 0-15 with a higher score being more indicative of depression.
Time Frame: 3 mo
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | 2 Growth Factors
Number analyzed (Participants) | 12
Units on a scale | 5 [0 to 12]

11. Secondary Outcome: Barthel Index
Description: Measure of disability in terms of performance of activities of daily living (ADL). The scores range from 0-100 with a higher score being associated with a higher level of independence.
Time Frame: 3 mo
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | 2 Growth Factors
Number analyzed (Participants) | 11
Units on a scale | 25 [0 to 100]

12. Secondary Outcome: Infarct Volume Using Anatomical MRI
Description: Measurement of infarct volume and percent change from baseline to Day 90.
Time Frame: 3 mo
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Beta-hCG + Erythropoietin
Number analyzed (Participants) | 7
percent change | -22 (34)

13. Secondary Outcome: Trail Making A Test
Description: Measure of memory and executive function where one is asked to connect dots consecutively based on the number of the dot. Test taker is allowed 2 minutes to connect the dots with a maximum score of 25 for all dots connected correctly.
Time Frame: 3 mo
Measure: Median (Full Range); unit: correct connections
Arm/Group | 2 Growth Factors
Number analyzed (Participants) | 7
correct connections | 8 [0 to 25]

14. Secondary Outcome: Trail Making B Test
Description: Measure of memory and executive function where one is asked to connect dots with letters and numbers alternating between number and letter and connecting dots consecutively. Test taker is allowed 4 minutes to connect the dots with a maximum score of 25 for all dots connected correctly.
Time Frame: 3 mo.
Measure: Median (Full Range); unit: correct connections
Arm/Group | 2 Growth Factors
Number analyzed (Participants) | 5
correct connections | 3 [0 to 11]

ADVERSE EVENTS:
Arm/Group | Beta-hCG + Erythropoietin
Serious Adverse Events (participants affected / at risk) | 6/15
Other Adverse Events (participants affected / at risk) | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Beta-hCG + Erythropoietin (N=15)
Death (General disorders) | 2 (2)
Deep Vein Thrombosis (Vascular disorders) | 2 (2)
Cerebral embolism (Nervous system disorders) | 1 (2)
Mediastinal sepsis (Infections and infestations) | 1 (1)
Retroperitoneal hemorrhage (General disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No